CLINICAL TRIAL: NCT02465216
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled, Clinical Trial to Evaluate the Safety and Immunogenicity of the ID93 + GLA-SE Vaccine in HIV Uninfected Adult TB Patients After Treatment Completion
Brief Title: Phase 2a ID93 + GLA-SE Vaccine Trial in TB Patients After Treatment Completion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Wellcome Trust (Other); South African Tuberculosis Vaccine Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IDRI-TBVPX-203
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; TB; Pulmonary; Vaccine; Adjuvant
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 2 mcg ID93 + 2 mcg GLA-SE Vaccine (Experimental): Two intramuscular injections of ID93 + GLA-SE at Days 0 and 56. Low dose of antigen and low dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 10 mcg ID93 + 2 mcg GLA-SE Vaccine (Experimental): Two intramuscular injections of ID93 + GLA-SE at Days 0 and 56. High dose of antigen and low dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE
- 2 mcg ID93 + 5 mcg GLA-SE Vaccine (Experimental): Two intramuscular injections of ID93 + GLA-SE at Days 0 and 56. Low dose of antigen and high dose of adjuvant. Placebo injection at Day 28 to maintain blind with the 3 dose arm.
  Interventions: Biological: ID93 + GLA-SE
- Placebo (Placebo Comparator): Two intramuscular injections of normal saline at Days 0 and 56, or Days 0, 28, and 56.
  Interventions: Other: Placebo
- 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 doses (Experimental): Three intramuscular injections of ID93 + GLA-SE at Days 0, 28, and 56. Low dose of antigen and high dose of adjuvant.
  Interventions: Biological: ID93 + GLA-SE

INTERVENTIONS:
Other: Placebo — Placebo
  Arms: Placebo
Biological: ID93 + GLA-SE — ID93 + GLA-SE
  Arms: 10 mcg ID93 + 2 mcg GLA-SE Vaccine; 2 mcg ID93 + 2 mcg GLA-SE Vaccine; 2 mcg ID93 + 5 mcg GLA-SE Vaccine; 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 doses

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of ID93 + GLA-SE vaccine when administered to adult pulmonary Tuberculosis (TB) patients, following successful completion of TB treatment with confirmed bacteriologic cure, in preparation for a future Phase 2b prevention of TB recurrence trial in the same population.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 to 60 years of age.
2. Subjects must have been successfully treated, i.e., completed the scheduled course of TB treatment as per the prevailing South African national guidelines, for MTB culture-confirmed, drug sensitive pulmonary TB, as evidenced by a record of positive liquid MTB culture with formal drug sensitivity testing (DST) and/or by Xpert MTB/RIF test at baseline.
3. Must have two separate samples showing bacteriologic confirmation of cure - defined in the first instance as Xpert MTB/RIF test negative, or, if Xpert MTB/RIF positive, as MTB liquid culture negative - on two successive occasions at least 30 days apart. Subjects who are sputum unproductive will be deemed Xpert MTB/RIF and MTB liquid culture negative.
4. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of each study injection, must not be breast-feeding, and be willing to avoid pregnancy for 3 months following first study injection. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide gel.
5. The following screening laboratory values must be within the laboratory reference range or, if abnormal, deemed not clinically significant and less than Grade 2 severity on the FDA Toxicity Scale, as determined by the PI and LMM or Sponsor Medical Advisor: ALT, AST, total bilirubin, creatinine, total WBC count, hemoglobin, and platelet count.
6. The HIV 1/2 antibody serology tests must be negative.
7. Must give informed consent, be able and willing to make all evaluation visits, be reachable by telephone or personal contact by the study site personnel, and be willing to remain in the study area for the duration of the trial.

Exclusion Criteria:

1. TB treatment failure, as evidenced by clinical diagnosis or a positive MTB liquid culture at month 4 or 5 after starting treatment. A positive MTB liquid culture at, or after, end of treatment would exclude subjects from receiving further study injections.
2. Previous course of TB treatment completed within 5 calendar years prior to obtaining baseline diagnostic sputum samples.
3. Receipt of any investigational products or investigational drug in the past 6 months or investigational vaccine ever.
4. Treatment with immunosuppressive drugs (e.g., oral or injected steroids, such as prednisone; high dose inhaled steroids) in the past 6 months. Topical steroids would be allowable.
5. Received incomplete or investigational, or non-standard TB drug regimen, other than the prevailing current South African national guideline as reference standard, or poor adherence to TB treatment regimen.
6. Diagnosed with rifampicin-resistant MTB strain (by Xpert MTB/RIF and/or culture and formal DST).
7. History of autoimmune disease or other causes of immunosuppressive states.
8. History or evidence of any acute or chronic illness (including diabetes mellitus, asthma), medical or surgical condition, or chronic heavy ethanol or drug use, or use of medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
9. Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines, eggs, or unknown allergens.
10. Subjects who are unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hatherill, MD, Principal Investigator — South African Tuberculosis Vaccine Initiative
Locations (3):
- South Africa (3):
  - TASK Applied Sciences, Cape Town
  - Desmond Tutu HIV Centre (DTHC), Cape Town
  - South African Tuberculosis Vaccine Initiative (SATVI), Worcester

REFERENCES:
- [Derived] Day TA, Penn-Nicholson A, Luabeya AKK, Fiore-Gartland A, Du Plessis N, Loxton AG, Vergara J, Rolf TA, Reid TD, Toefy A, Shenje J, Geldenhuys H, Tameris M, Mabwe S, Bilek N, Bekker LG, Diacon A, Walzl G, Ashman J, Frevol A, Sagawa ZK, Lindestam Arlehamn C, Sette A, Reed SG, Coler RN, Scriba TJ, Hatherill M; TBVPX-203 study team. Safety and immunogenicity of the adjunct therapeutic vaccine ID93 + GLA-SE in adults who have completed treatment for tuberculosis: a randomised, double-blind, placebo-controlled, phase 2a trial. Lancet Respir Med. 2021 Apr;9(4):373-386. doi: 10.1016/S2213-2600(20)30319-2. Epub 2020 Dec 8. PMID 33306991

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2 mcg ID93 + 2 mcg GLA-SE Vaccine | 10 mcg ID93 + 2 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 Doses | Placebo
Started | 15 | 5 | 14 | 14 | 12
Completed | 12 | 5 | 13 | 12 | 9
Not Completed | 3 | 0 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 mcg ID93 + 2 mcg GLA-SE Vaccine | 10 mcg ID93 + 2 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 Doses | Placebo | Total
Number analyzed (Participants) | 15 | 5 | 14 | 14 | 12 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 5 | 14 | 14 | 12 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 7 | 2 | 4 | 27
  Male | 4 | 2 | 7 | 12 | 8 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Mixed Race | 10 | 1 | 11 | 7 | 8 | 37
  Black African | 5 | 4 | 3 | 7 | 4 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 15 | 5 | 14 | 14 | 12 | 60
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.6 (2.32) | 22.8 (5.4) | 19.6 (2.38) | 21.4 (4.92) | 21.4 (1.94) | 20.9 (3.39)

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Safety outcomes will include solicited adverse events within 7 days and unsolicited adverse events within 28 days after each study injection; and serious adverse events after the first study injection until end of study follow-up.
Time Frame: 224 days
Measure: Number; unit: participants
Arm/Group | 2 mcg ID93 + 2 mcg GLA-SE Vaccine | 10 mcg ID93 + 2 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 Doses | Placebo
Number analyzed (Participants) | 15 | 5 | 14 | 14 | 12
participants
  Local Injection Site Reactions | 5 | 4 | 10 | 8 | 3
  Solicited Systemic Reactions | 1 | 0 | 1 | 1 | 0
  Any Adverse Event | 12 | 5 | 13 | 12 | 9
  Serious Adverse Events | 0 | 0 | 0 | 0 | 2

2. Secondary Outcome: Immunogenicity Responder Rate
Description: Immunogenicity will be evaluated by measuring humoral and cellular responses to ID93 + GLA-SE at Day 70.
Time Frame: Day 70
Population: Those participants without major protocol deviations and with samples available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mcg ID93 + 2 mcg GLA-SE Vaccine | 10 mcg ID93 + 2 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 Doses | Placebo
Number analyzed (Participants) | 13 | 5 | 13 | 11 | 11
Participants
  IgG antibody responder rate: number analyzed (Participants) | 12 | 5 | 13 | 11 | 11
  IgG antibody responder rate | 12 | 5 | 13 | 11 | 0
  CD4 T cell responder rate (whole antigen stim): number analyzed (Participants) | 13 | 5 | 11 | 9 | 10
  CD4 T cell responder rate (whole antigen stim) | 4 | 2 | 10 | 1 | 1

ADVERSE EVENTS:
Time Frame: 224 days
Arm/Group | 2 mcg ID93 + 2 mcg GLA-SE Vaccine | 10 mcg ID93 + 2 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine | 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 Doses | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5 | 0/14 | 0/14 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/14 | 0/14 | 2/12
Other Adverse Events (participants affected / at risk) | 12/15 | 5/5 | 13/14 | 12/14 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mcg ID93 + 2 mcg GLA-SE Vaccine (N=15) | 10 mcg ID93 + 2 mcg GLA-SE Vaccine (N=5) | 2 mcg ID93 + 5 mcg GLA-SE Vaccine (N=14) | 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 Doses (N=14) | Placebo (N=12)
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium tremens (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mcg ID93 + 2 mcg GLA-SE Vaccine (N=15) | 10 mcg ID93 + 2 mcg GLA-SE Vaccine (N=5) | 2 mcg ID93 + 5 mcg GLA-SE Vaccine (N=14) | 2 mcg ID93 + 5 mcg GLA-SE Vaccine 3 Doses (N=14) | Placebo (N=12)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 3 (4) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 5 (6) | 4 (4) | 10 (16) | 7 (13) | 3 (3)
ALT increased (Investigations) | 2 | 0 | 1 | 3 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1 | 1 | 0 | 0
WBC count decreased (Investigations) | 0 | 1 | 2 | 2 | 0
WBC count increased (Investigations) | 1 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 0 | 3
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Tonsilitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0
URTI (Infections and infestations) | 3 | 1 | 3 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No